CLINICAL TRIAL: NCT06285344
Title: The Impact of Individual Workload and Fatigue Levels on Sleep Perception in Operating Room Nurses: A Multicenter Cross-Sectional and Correlational Study
Brief Title: Impact of Workload and Fatigue on Sleep in OR Nurses
Status: Not yet recruiting | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Researcher Asisstan, Kilis 7 Aralik University
Other Study IDs: kilis_3
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Shift Work; Sleep Perception
Keywords: Operating Room Nurses; Workload; Fatigue; Sleep Quality; Patient Safety; Healthcare Professionals; Stress Levels; Shift Work; Sleep Perception; Nurse Well-being; Surgical Settings; Emotional Challenges; Patient Care Quality
MeSH Terms: conditions — Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the impact of individual workload and fatigue levels on the sleep quality of operating room (OR) nurses, highlighting a critical aspect of healthcare professionals' well-being that directly affects patient safety and care quality. Operating room nurses face unique challenges due to the high-stress, fast-paced environment of surgical settings, which can lead to increased stress levels, emotional challenges, and a higher incidence of fatigue compared to other nursing specialties. Factors contributing to this fatigue include the demanding nature of surgical procedures, the need for constant vigilance, and the irregular hours associated with shift work, all of which can impair sleep quality.

The literature review suggests that while the relationship between workload, fatigue, and sleep quality has been extensively studied in general nursing populations, there is a lack of specific focus on operating room nurses. These professionals work under distinct conditions that may exacerbate the effects of workload and fatigue on sleep quality, yet comprehensive studies targeting this group are limited. Understanding the nuances of how workload and fatigue specifically impact the sleep quality of OR nurses is crucial for developing targeted interventions aimed at improving their health and job performance, thereby enhancing patient care and safety.

This cross-sectional and correlational study seeks to fill the gap in the literature by examining the specific effects of workload and fatigue on sleep perception among OR nurses. By identifying these relationships, the study aims to contribute valuable insights into strategies for mitigating fatigue and improving sleep among this critical group of healthcare workers, with the ultimate goal of ensuring both nurse well-being and patient safety.

DETAILED DESCRIPTION:
Operating room nurses play a critical role in surgical environments (Aorn 2020). The intense pace of the operating room environment can expose nurses to high workloads, increased stress levels, and emotional challenges (Alrawashdeh H 2021) (Teymoori, E 2022). The continuously changing and complex structure of modern healthcare services can further deepen these effects. Specifically, emergencies or unexpected complications during surgery can expose operating room nurses to different stress factors compared to other nurses (Teymoori, E 2022). The intense work environment of operating room nurses subjects them to high workloads and stressors, leading to stress and fatigue due to various factors (Jang 2021; Yuan SC 2011, Fang 2008, Shahzad, 2021). Fatigue represents a reduction in physical and emotional energy, a lack of motivation, and a general sense of exhaustion. Fatigue in nurses has been associated with factors such as high workloads, inadequate workplace support, challenging physical conditions, and shift work (Khande 2017). Particularly, day and night shifts can lead to increased workloads and consequently to higher rates of anxiety and depression (Warren 2008, Jang 2021 Barker 2011 Smith-Miller 2018 Clendon J 2019 Rathore H 2012 Yang YH 2012 Lee EJ 2014). This situation can lead to acute or chronic fatigue and even negative cycles (Barker LM 2011, Kawano 2008).

Workload is one of the biggest challenges faced by operating room nurses. The perception of workload among nurses can negatively affect their levels of fatigue, which in turn can reduce sleep quality (Cho, H. 2022; Dong 2017; Liu, Y., 2022). High workload can deplete nurses' physical and emotional energies (Akansel 2019)(Fan, 2021; Ghasemi,2019), leading to increased levels of fatigue. It can also negatively affect their decision-making abilities during critical surgical procedures. Moreover, high levels of fatigue can reduce the quality of care provided by nurses to patients, leading to negative effects on patient safety and treatment outcomes (Cho 2022)(Cho, H. 2022) (Dong 2017)(Metthevs 2011) (Liu, Y., 2022) and thus can affect sleep quality (Lin 2014).

Sleep quality is a critical factor for the overall health and job performance of operating room nurses. Generally, among health professionals, the primary causes of fatigue include circadian rhythm sleep disorders and sleep deprivation (Garrubba 2019, Jang 2021) Insomnia not only causes fatigue in nurses but can also negatively affect their psychomotor skills, reduce motivation and job performance, and impair their ability to maintain safe workplace behaviors (Dong 2017, Warren 2008, Choi UE 2016 Seol2018) This situation can lead to errors in procedures performed on patients and even harm to themselves [^8,Huckels-Baumgart, S.,2017) (Jones, T.2014) (Minnick, A 2012) (Pugh, C. 2011). Therefore, fatigue in operating room nurses not only affects them but also directly impacts patient safety and care quality (Garrubba 2019, Jang 2021) Preventing fatigue and eliminating the adverse conditions resulting from fatigue are essential for the safety of both patients and healthcare workers (Warren 2008, Smith-Miller 2014).

The effects of workload and fatigue levels on sleep quality among operating room nurses are significant issues for the nurses' overall health and job performance. The literature extensively examines the relationship between workload, fatigue, and sleep quality (Fan, 2021; Ghasemi,2019). Specifically, understanding the fatigue levels of operating room nurses is vital for the safety and health of both patients and nurses (Yamin 2020; Gurses 2009). The relationship between workload perception and sleep quality is critical for optimizing nurses' clinical performance and patients' health outcomes (Metthevs 2011). It has been indicated that a high perception of workload can have negative effects on fatigue and sleep quality.

The literature generally focuses on the general nurse population and has not sufficiently examined the demographic characteristics of operating room nurses and the potential effects of these characteristics on workload perception, fatigue, and sleep quality. Moreover, comprehensive studies specifically focusing on this topic are limited. The unique working conditions of operating room nurses, and the relationship between workload perception, fatigue, and sleep quality, should be examined more specifically and in detail. The findings obtained will contribute to the development of strategies to reduce fatigue among operating room nurses and improve their perception of sleep. This study will be conducted with the aim of determining the impact of individual workload and fatigue levels on sleep perception among operating room nurses and identifying the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who have been working as operating room nurses in the hospitals where the study is conducted for at least one year,
* Nurses who are willing to participate in the study will be included.

Exclusion Criteria:

* Data from nurses who wish to withdraw from the study at any stage will be excluded from the research.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study focuses on operating room (OR) nurses with at least one year of experience in various hospitals. These participants are chosen for their specialized knowledge in the surgical environment, ensuring they provide insights into workload, fatigue, and sleep quality. Inclusion is based on voluntary consent, aiming to collect data from a group well-versed in the unique challenges and stressors of OR settings. This demographic is particularly valuable for exploring how their demanding roles affect sleep and well-being.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Demographic Information Form | up to 12 weeks
  This form gathers nurses' demographic details through seven multiple-choice questions, covering aspects like age, gender, marital status, nursing experience, operating room nursing experience, chronic conditions, and regular medication usage.
Individual Workload Perception Scale (IWPS) | up to 12 weeks
  Initially developed in 2003 by Cox and colleagues and later adapted to Turkish in 2011 by Saygılı and Çelik, the IWPS assesses workload perception with a reliability coefficient of 0.894. It comprises 31 items across five categories: Supervisor Support, Colleague Support, Unit Support, Work Environment Workload Features, and Job Sustainability. Scoring is done on a 5-point Likert scale, with total scores ranging from 31 to 155, where higher scores suggest a more positive perception of workload.
Chalder Fatigue Scale (CFS) | up to 12 weeks
  The CFS, developed by Chalder et al. in 1993 and revised in 2010, is designed to measure fatigue levels. It includes two subscales for Physical and Mental Fatigue, with reliability ranging from 0.72 to 0.87. The scale consists of 11 items, which can be scored using either a bi-modal (0-1) or a 4-point Likert scale (0-3), with higher scores indicating greater fatigue levels.
Richard-Campbell Sleep Questionnaire (RCSQ) | up to 12 weeks
  Developed in 1987 by Richards, the RCSQ aims to evaluate different aspects of sleep quality using 6 items scored on a scale from 0 to 100. The Turkish version's reliability, assessed by Karaman Özlü and Özer in 2015, stands at 0.91. Higher scores on this scale denote better sleep quality, with detailed scoring ranges indicating varying levels of sleep quality from very poor to excellent.

CONTACTS AND LOCATIONS:
Overall Officials: islam elagöz, MsC, Study Director — devlet hastanesi
Locations (1):
- Islam Elagöz, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan ensures confidentiality and ethical compliance, using a secure, anonymized database for data access by verified researchers post-publication. Key aspects include anonymization, controlled access, a data use agreement, a sharing timeline, supporting documentation, and ethical oversight. This strategy balances scientific advancement with participant privacy.